CLINICAL TRIAL: NCT05440526
Title: Efficacy of the Mini-plate Anchored Herbst Appliance Versus the Dentally Anchored Fixed Functional Appliance in Young Adult Class II Orthodontic Patients; A Randomized Clinical Trial
Brief Title: the Mini-plate Anchored Herbst Appliance Versus the Dentally Anchored Fixed Functional Appliance
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mahmoud M. Fathy Aboelmahasen, Clinical professor of orthodontics - Faculty of dental medicine, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 586/307
Record Dates: First submitted 2022-06-27; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Class II Malocclusion
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Herbst Group (Active Comparator): • Group I: Include ten young adult orthodontic patients who are treated by using fixed orthodontic appliances followed by the type IV Herbst appliance (mini plate anchored appliance). The age of patients will be (18-20y).
  Interventions: Procedure: Herbst Group
- TFBC Group (Active Comparator): • Group II: Include ten young adult orthodontic patients who are treated by using fixed orthodontic appliances followed by the Twin Force Bite Corrector appliance (dentally anchored appliance). The age of patients will be (18-20y).
  Interventions: Device: TFBC Group

INTERVENTIONS:
Procedure: Herbst Group — Herbst Group:
  1. Two mini plates are chosen, the last hole in every plate is used to solder the ball housing of type IV Herbst appliance.
  2. The two mini plates are placed bilateral at the mandibular symphysis and fixed by at least 3 screws, the surgical wound is sutured.
  3. The surgical wound is left for 2 weeks for proper soft tissue healing, in the meantime separation in the arch, band placement on the first premolar and molar bilateral followed by impression for construction of the upper Herbst splint.
  Arms: Herbst Group
Device: TFBC Group — TFBC Group:
  1. The patients will be treated by fixed orthodontic appliance with using series of orthodontic NiTi arch wires for levelling and alignment.
  2. Installation of series of orthodontic stainless steel arch wires until 0.0019 x 0.0025 inch for both arches.
  3. Installation of the Twin Force Bite Corrector appliance for 4 to 6 months.
  4. Using of class ΙΙ intra-oral elastics for both sides for 2 to 3 months.
  Arms: TFBC Group

SUMMARY:
the objective of the current study is to compare the dentofacial effects of the mini-plate anchored Herbst appliance Versus the dentally anchored Twin force bite corrector Appliance in Young Adult Class II Orthodontic Patients with retruded mandible.

DETAILED DESCRIPTION:
Study design:

Prospective randomized clinical study.

Study setting and population:

This study will be conducted on twenty orthodontic patients. The number of patients was dependent on a power study.

Sample size calculation was based on the observed average effect size derived from previous article addressing "the effect of skeletally anchored Forsus FRD using miniplates for the treatment of Class II malocclusion.

Intervention:

The orthodontic patients involved in this study will be treated by using fixed orthodontic appliances followed by one of two different types of fixed functional appliances; the type IV Herbst appliance (miniplate anchored appliance) and the Twin Force Bite Corrector (dentally anchored appliance). According to the type of the fixed functional appliance the patients will be randomly divided into two groups. The random allocation will be achieved by computer software:

* Group I: Include ten young adult orthodontic patients who are treated by using fixed orthodontic appliances followed by the type IV Herbst appliance (mini plate anchored appliance). The age of patients will be (15-20y).
* Group II: Include ten young adult orthodontic patients who are treated by using fixed orthodontic appliances followed by the Twin Force Bite Corrector appliance (dentally anchored appliance). The age of patients will be (15-20y).

Records:

The following diagnostic records will be taken for each patient before and after the fixed functional orthopedic treatment:

1. Standardized study casts.
2. Standardized extra-oral and intra-oral photographs.
3. Lateral cephalometric and panoramic radiographs.

Treatment steps:

As for Group Ι:

1. Two mini plates are chosen, the last hole in every plate is used to solder the ball housing of type IV Herbst appliance.
2. The two mini plates are placed bilateral at the mandibular symphysis and fixed by at least 3 screws, the surgical wound is sutured leaving an extended part of the plate in the oral cavity which contain the soldered ball housing.
3. The surgical wound is left for 2 weeks for proper soft tissue healing, in the meantime separation in the arch, band placement on the first premolar and molar bilateral followed by impression for construction of the upper Herbst splint.
4. Cementation of upper Herbst splint with connecting the telescopic piston through fitting of the plunger into the tube bilaterally.
5. When reactivation of the telescopic piston is needed, extension rings are used.

As for Group ΙΙ:

1. The patients will be treated by fixed orthodontic appliance with using series of orthodontic NiTi arch wires for levelling and alignment.
2. Installation of series of orthodontic stainless steel arch wires until 0.0019 x 0.0025 inch for both arches.
3. Installation of the Twin Force Bite Corrector appliance for 4 to 6 months.
4. Using of class ΙΙ intra-oral elastics for both sides for 2 to 3 months.
5. Finally follow finishing steps for each patient.

Data management and analysis:

The collected data will be tabulated statistically analyzed using Statistical Package for Social Sciences (SPSS, version 18, Inc, and Chicago, Ill).

ELIGIBILITY:
Inclusion Criteria:

* Participants will be selected based on the following inclusion criteria:

  1. Skeletal class 2 malocclusion due to mandibular retrusion with increased overjet (SNA= 82±4, ANB=≥4°).
  2. Mandibular arch with minimum (up to 4mm) or no crowding.
  3. All permanent teeth are erupted (3rd molar not included).
  4. Good oral and general health.
  5. No systemic disease or regular medication that could interfere and/or affect orthodontic teeth movement.
  6. No previous orthodontic treatment.

Exclusion Criteria:

- 1. Patients with a blocked-out tooth that will not allow for placement of the bracket at the initial bonding appointment.

2. Patients with untreated decay or any endodontic lesions.

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Amount of changes in dentoskeletal cephalometric measurements between Herbst Group and TFBC group | one year and four months
  lateral cephalometric radiograph was analysed by dolphin software to assess the following angular (in degree) and linear (in mellimeter) measurements : SNA - SNB - ANB - Y AXIS angle - facial angle - (co - A) - (co - gn) - ( upper 1 - SN) - (lower 1 - MP) - overjet - over bite - soft tissue convexity angle.

SECONDARY OUTCOMES:
Amount of changes in dentoskeletal cephalometric measurements within each group separately | one year and four months
  lateral cephalometric radiograph was analysed by dolphin software to assess the following angular (in degree) and linear (in mellimeter) measurements : SNA - SNB - ANB - Y AXIS angle - facial angle - (co - A) - (co - gn) - ( upper 1 - SN) - (lower 1 - MP) - overjet - over bite - soft tissue convexity angle.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M. Fathy Aboelmahasen, PHD, Principal Investigator — Lecturer of orthodontics - Faculty of dental medicine - Al-Azhar university
Locations (1):
- Nasr city, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No